CLINICAL TRIAL: NCT02266316
Title: A Randomised Controlled Trial of an Air Warming Mask to Increase Exercise Tolerance in Patients With Stable and Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Use of an Air Warming Mask for Exercise in Patients With COPD V1.0
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: WARM/COPD/1112
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mask (Experimental): Using mask that warms air at the mouth by utilising body heat
  Interventions: Device: Air warming mask
- No mask (No Intervention): Not using any mask that warms air at the mouth by utilising body heat

INTERVENTIONS:
Device: Air warming mask — Mask that warms air at the mouth
  Arms: Mask

SUMMARY:
The World Health Organisation defines chronic obstructive pulmonary disease (COPD) as 'not one single disease but an umbrella term used to describe chronic lung diseases that cause limitations in lung airflow' covering emphysema and chronic bronchitis; and estimates (2004) that worldwide there are currently 64 million sufferers with 3 to 4 million in the UK.

COPD results from damaged airways in the lungs, causing them to become narrower and making it harder for air to get in and out of the lungs. It is diagnosed by measuring the amount of air that can be expelled in the first second of breathing out (FEV1) in litres per second.

COPD is a progressive disease and the condition can have a serious impact on the quality of life of sufferers. Going out in very cold weather can cause an immediate drop in FEV1, and increased breathlessness.

This is a randomised crossover controlled trial of participants with COPD. It compares the effectiveness of an air-warming face mask which covers the mouth compared with no face covering, in increasing participants exercise capacity and quality of life in cold weather. The mask warms air at the mouth by drawing on air warmed beneath the participants clothing, through a 20cm long hollow plastic tube and a one-way inspiratory valve into the mask. Air is expired through the nose.

24 participants with moderate or severe COPD, will undertake 3 exercise tests on 3 separate days. Two tests will be in an environmentally controlled chamber performed at 5°C with participants wearing either the mask or no face covering. The third test will be performed at ambient temperature outside the chamber.

The order will be determined by random allocation. Participants will undergo the Treadmill 6 Minute Walk Test; various measurements will be taken, all of which will be non-invasive.

DETAILED DESCRIPTION:
Purpose and design

Previous studies have demonstrated the detrimental effect of inhaled cold air for COPD sufferers [1].

Recommendations for COPD sufferers suggest covering the mouth or mouth and nose during cold weather to reduce the impact of cold air, but to date there is no information about how effective this actually is. A previous study of an alternative mask only involved 9 participants with moderate levels of COPD [2].

A further study is needed to establish how effective masks are during cold conditions as they could be a simple, inexpensive way of improving quality of life through exercise, further deterioration of the condition can result from sufferers becoming more sedentary.. A better understanding could be useful for clinicians to advise patients on how and why they can protect themselves from the cold.

NICE guidelines published in 2004 and 2010 highlight the importance of pulmonary rehabilitation in improving the quality of life of COPD patients incorporating a programme of physical training, disease education, nutritional, psychological and behavioural intervention. Exercise has many health benefits, including reducing depression and anxiety; clinical depression and anxiety are common problems for participants with COPD. Exercise can be, or perceived to be difficult for COPD sufferers during cold periods due to brochoconstriction (constriction of the airways in the lungs) and many sufferers can be confined indoors during cold weather in the winter months.

The primary aim of the study is to answer the question of whether a face mask, which provides air warmed by the body and brought to the mouth, increases exercise capacity in participants with stable and moderate or severe COPD, during cold weather. Cold weather can cause an immediate drop in FEV1 and increased breathlessness discouraging sufferers from going outdoors during the winter.

The sample size of 24 participants has been determined from a power calculation by the trial statistician.

The study has been designed as a crossover trial, with each participants performing an exercise test three times. The first test will be performed in ambient temperature with no face covering. Participants will have their health assessed and be trained on how to use a treadmill. The other two tests will be performed in a climate controlled chamber set at 5oC, once wearing the test mask and once wearing no mask or face covering. The order of these two tests will be determined at random by the statistician. The participants will dress as they feel appropriate for a cold winter's day except for any scarf or muffler.

The study will be held in the spring or autumn to avoid periods of cold weather but also to avoid the hot summer months as excessive heat can equally trigger increased breathlessness in COPD sufferers.

The effects of exercise and exercise tolerance testing on COPD participants has been researched and documented elsewhere and is not the purpose of this study [3] so participants will not undergo rigorous exercise patterns such as the full Bruce Protocol[4] (standardised protocol that monitors functions in exercising participants). The American Thoracic Society has produced a protocol for the Six-Minute Walk Test which is a simple test measuring the distance a patient can walk on a hard flat surface in a period of 6 minutes (6MWD)[5]. The 6-minute walk test (6MWT) is commonly used to assess changes in functional exercise capacity in COPD participants following pulmonary rehabilitation with the primary outcome reported being the distance walked during the test. Studies have shown that the 6MWT can be equally used on a treadmill [6]. The choice of protocol was made after consultation with a respiratory clinician and a sports physiologist.

The mask is a simple device comprising a plastic face mask (with elastic strap) and plastic tube that feeds into it with a one way valve to prevent moisture laden breath returning down the tube. The wearer inserts the tube into their own clothing and inhales air preheated by their own body. The device is made of medically approved, flexible plastics. The wearer inhales through the mouth and exhales through the nose. The shape and size of the mask has been determined by research conducted by the Health Design & Technology Institute based at Coventry University and it is configured to fit the majority of participants of any gender or ethnicity. The material chosen is one which is of a softness which is sufficiently firm to maintain shape whilst sufficiently soft to be comfortable worn next to the skin.

Participants will undertake three tests on three separate visits. The first test will comprise of walking for 6 minutes on a treadmill in ambient temperature wearing appropriate clothing and no mask. The other two tests will comprise of once walking for 6 minutes on a treadmill inside the environment chamber, with the temperature set to 5oC wearing the warm air mask and once walking for 6 minutes on a treadmill inside the environment chamber, with the temperature set to 5oC but not wearing any face covering. The order of these two tests for each participants will be determined at random by the trial statistician.

Pulmonary function will be assessed immediately before and after the exercise test using a spirometer. This will measure airflow obstruction by measuring the forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) (the total amount of air that you expire in one breath in litres per second). Both measurements are predictive of COPD and it would be expected that FEV1 would decrease when a COPD sufferer breathes in cold air.

Participants will also be asked to provide a rating on the Perceived Exertion Scale (ranks from 1 to 10) and breathlessness on the Borg scale during the exercise test (ranks from 1 to 10 with a written description of each level). If participants rank their breathlessness above 5 (severe breathlessness) the exercise test will be stopped immediately. Oxygen saturation and heart rate will be continuously monitored during the exercise tests.

At the end of each exercise test, participants will have a rest period during which time they will be monitored by a clinician. Full resuscitation facilities will be available including defibrillator.

1. Kosela H, Pihlajamaki J, Pekkarinene H, Tukiainen, H O (1998) Effect of cold air on exercise capacity in COPD: Increase or decrease? Chest 113: 1560-1565.
2. Seifer J G The Cardiopulmonary effect of a heat and moisture exchange mask on COPD patients during cold exposure. Presented at the European Respiratory Society Annual Congress, Vienna 2009
3. Cooper, C. B. Exercise in chronic pulmonary disease: aerobic exercise prescription. Med. Sci. Sports Exerc., Vol. 33, No. 7, Suppl., pp. S671-S679, 2001.
4. Bruce et al Normal Respiratory and circulatory pathways of adaptation in exercise J Clin Invest. 1949 November; 28(6 Pt 2): 1423-1430
5. ATS statement: Guidelines for the Six-Minute Walk Test. Am J Respir Crit Care Med Vol 166 pp111-117, 2002
6. Almeida et al, Hallway versus treadmill 6 minute Walk Tests in Patients with Chronic Obstructive Pulmonary Disease. Respiratory Care December 2009 Vol54 No 12

ELIGIBILITY:
Inclusion Criteria:

* Males or females diagnosed with COPD, GOLD stage 2 to stage 4
* Stable COPD
* ≥40 years old
* Ability to walk for 6 minutes without stopping
* Medical Research Council (MRC) scale of dyspnoea - grade 3 or above (grade 3 means a patient is limited to walking slower than contemporaries on the level because of breathlessness, or has to stop for breath when walking at own pace).

Exclusion Criteria:

* Significant disease other than COPD
* Ischaemic heart disease
* Use of supplemental oxygen therapy
* Participants who are unable to walk
* Unstable or life-threatening cardiac arrhythmia
* History of myocardial infarction
* Cold, flu like illness, or other chest infection in the last 8 weeks
* Participants who are currently experiencing an exacerbation of their COPD
* Participants who have experienced an exacerbation in the previous 8 weeks
* Participants who have a known reaction to medical plastics

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure for the study is the difference between forced expiratory volume in one second (FEV1) in litres per second before and after a 6 minute walk. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Roy Kennedy, PhD, Principal Investigator — University of Worcester
Locations (1):
- University of Worcester, Worcester, Worcestershire, United Kingdom